CLINICAL TRIAL: NCT02944942
Title: Risk Factors for Postoperative Nausea/Vomiting After Implementation of Prophylaxis Guideline for High Risk Patients
Brief Title: Risk Factors for Postoperative Nausea/Vomiting
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Other Study IDs: HE571413
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postoperative nausea and vomiting: Group 1: Patients undergoing general anesthesia with postoperative nausea and vomiting Group 2: Patients undergoing general anesthesia without postoperative nausea and vomiting
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: General anesthesia — Patients undergoing general anesthesia

SUMMARY:
General anesthetic technique plays a key role in most surgical procedures. This technique has some complications especially postoperative nausea/vomiting (PONV). This complication can lead to serious problems. Department of Anesthesiology has developed and implemented a PONV prophylaxis guideline for high risk PONV patients but PONV still remains.

DETAILED DESCRIPTION:
Objective: To identify risk factors for PONV after implementation of PONV prophylaxis guideline.

Methods: This will be a retrospective analytic study. Relevant clinical data from medical records of adult patients undergoing general anesthesia in Srinagarind Hospital from November 2014 to February 2015 will be used to identify relevant risk factors.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-III

Exclusion Criteria:

* Incomplete or illegible medical records
* Patients who underwent cardio-thoracic surgery
* Patient who had chronic treatment with antiemetic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | through study completion, an average of 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (1):
- Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Result] Blanc VF, Ruest P, Milot J, Jacob JL, Tang A. Antiemetic prophylaxis with promethazine or droperidol in paediatric outpatient strabismus surgery. Can J Anaesth. 1991 Jan;38(1):54-60. doi: 10.1007/BF03009164. PMID 1989740
- [Result] Chatterjee S, Rudra A, Sengupta S. Current concepts in the management of postoperative nausea and vomiting. Anesthesiol Res Pract. 2011;2011:748031. doi: 10.1155/2011/748031. Epub 2011 Nov 3. PMID 22110499
- [Result] Doubravska L, Dostalova K, Fritscherova S, Zapletalova J, Adamus M. Incidence of postoperative nausea and vomiting in patients at a university hospital. Where are we today? Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2010 Mar;154(1):69-76. doi: 10.5507/bp.2010.012. PMID 20445713
- [Result] Jokinen J, Smith AF, Roewer N, Eberhart LH, Kranke P. Management of postoperative nausea and vomiting: how to deal with refractory PONV. Anesthesiol Clin. 2012 Sep;30(3):481-93. doi: 10.1016/j.anclin.2012.07.003. Epub 2012 Aug 14. PMID 22989590